CLINICAL TRIAL: NCT04534361
Title: "Dimensional Hard Tissue Changes Resulted at Removed Peri-implantitis Implant Sites: A Retrospective Study".
Brief Title: Alveolar Ridge Sequelae Due to Peri-implantitis: a Retrospective Observational Study
Status: Completed | Type: Observational
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Ramón Pons Calabuig, Dentistry, Master in Periodontics and Implants, Universitat Internacional de Catalunya
Other Study IDs: SES-CEI-120820
Record Dates: First submitted 2020-08-26; First posted 2020-09-01 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Dental Implant; Peri-Implantitis; Bone Remodeling
Keywords: dental implant; dental implant failure; peri-implantitis; bone loss; bone remodeling; implant explantation
MeSH Terms: conditions — Peri-Implantitis; Bone Diseases, Metabolic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: CBCT measurements — No intervention will be performed on patients for this study. Based on the CBCTs already done previously of the patients in the sample, linear measurements will be taken in order to assess dimensional changes of the alveolar ridge at 1, 3, 5 and 7 mm from the bone crest in the CBCTs taken before and after implant explantation, 4-6 months apart.

SUMMARY:
The scientific evidence available at present regarding the alterations suffered by the alveolar ridge after the explantation of implants that have been considered to be abandoned due to periimplantitis, as well as the remaining sequelae from said treatment, is scarce and inconclusive.

Regarding this background, it is speculated that the different types of peri-implant defects present different bone remodeling and different sequelae after the explantation of the implants affected by peri-implantitis.

Thus, it has been hypothesized that the peri-implant defect configuration has an influence on the radiographic bone alterations that occur after explantation.

In order to test this hypothesis, a retrospective study has been designed as it follows: Patients who have undergone implant placement procedure and suffer from peri-implantitis will be consecutively included in the study. In addition, patients should present at least 2 CBCTs taken before and after explantation, 4-6 months apart. Linear measurements will be taken in order to assess dimensional changes of the alveolar ridge at 1, 3, 5 and 7 mm from the bone crest.

DETAILED DESCRIPTION:
Peri-implant diseases have been a growing problem for the last decades. A recent cross-sectional study conducted in the Spanish population has shown a prevalence of mucositis and peri-implantitis at the implant level of 27% and 20%, and of 27% and 18% at the patient level, respectively (Rodrigo et al. 2018). As the peri-implant disease progresses, it has been observed that it generates different types of defects around implants affected by this pathology. Recently, Monje et al. 2019, have classified these defects according to their morphology (infrabony defects, supracrestal/horizontal defects or combined defects) and according to the depth of the defect and total bone loss/total implant length (3-4mm/<25% of implant length, 4-5mm/≥25-50% of implant length, >6mm/>50% of implant length (Monje et al. 2019).

Bone remodeling, as well as the sequelae or morphological alterations suffered by the alveolar ridge after tooth extraction have been widely described in the literature (Amler et al. 1960, Evian et al. 1982, Cardaropoli et al. 2003). In an animal model, Araujo and coworkers described the alterations of the alveolar ridge following tooth extraction; observing that bone height reduction of the buccal plate was more pronounced than the lingual, and that vertical bone loss was always associated with horizontal bone loss (Araujo et al. 2005). In contrast, the evidence available nowadays regarding the alterations suffered by the alveolar ridge after the explantation of implants that have been considered to be removed due to peri-implantitis, as well as the remaining sequelae from said treatment, is scarce and inconclusive.

Therefore, the the primary objective of this study will be to evaluate radiographically the influence of the peri-implant defect configuration on the radiographic bone alterations after implant explanation.

In this sense, a retrospective observational study will be design. The protocol of which will be approved by the Ethics Committee of the University of Extremadura (Badajoz, Spain), and will follow the Declaration of Helsinki on human studies. In addition, this study will be reported in accordance with the Analysis Strenghtening the Reporting of Observational Studies in Epidemiology (STROBE) Statement .

Patient recruitment will be obtained from a private practice exclusively dedicated to periodontics and implantology. Edentulous patients, either total or partial, who previously underwent implant placement procedure will be consecutively included in the study. A prerequisite for being eligible for the study was to have at least 2 CBCts, one taken before explantation in order to diagnose peri-implantitis; and the other taken after explantation.

In order to define a peri-implantitis case, it will be based on the consensus report of Workgroup 4 of the 2017 World Workshop on the Classification of Periodontal and Peri-implant Diseases and Conditions (Berglundh et al., 2018), in which it was stated that, in the absence of baseline information, the diagnosis of peri-implantitis required: presence of bleeding and/or suppuration on gentle probing, probing depth ≥6 mm and bone level ≥3mm apical to the most coronal portion of the implant or at the rough-smooth interface in transmucosal implants.

Once defined, several variables will be recorded, including both patient- and implant-related ones. The former will include age, gender, type of edentulism (total/partial), history of periodontal disease (mild, moderate or severe), tobacco smoking (heavy smoker >10 cigarettes/day; light smoker <10 cigarettes/day, former smoker 0 cigarette/day or non-smoker), numbers of implant per patient, and keratinized mucosa (0, <2 or ≥2 mm). Implant-related variables will include position (mandible / maxilla / anterior / posterior), implant system (brand, diameter, length and type of connection), implant macrodesign (transmucosal/bone level), type of prosthesis (single/multiple; screw/cement-retained), as well as explantation method (trephine, tweezers, forceps or implant removal kit). In addition, whether regeneration was performed or not after explantation will be recorded, as well as the material used for it.

For the radiographic assessment, images were acquired by CBCT i-CAT Model 17-19 (Imaging Sciences International LLC, Hatfield, PA, USA). The imaging parameters were set at a width and depth of 16 × 13 mm, 120 kVp, 20.27 mAs, scan time 14.7 seconds, resolution 0.25 voxel and a field of view (FOV), which varied based on the scanned region. Defect morphology and severity were determined using the OnDemand3D software (Cybermed, Seoul, Korea) by one previously calibrated examiner.

Prior to the assessment of the different radiographic variables, two reference lines will be established: longitudinal axis of the implant and a perpendicular line to it tangent to a reference point (sinus floor in the maxilla and mandibular base in the mandible). Several parameters will be assessed before and after explantation in each implant, including: bone-to-implant contact (BIC) at 4 sites (mesial, distal, buccal, lingual), defined as the first contact between the bone and the implant surface, assessed from the most coronal part of the intraosseous component of the implant; bone plate thickness (BPT), assessed at buccal and lingual in mm. The reference point will be the bone crest and bone thickness will be recorded at 1, 3, 5 and 7 mm from the crest. In addition, ridge width (RW) will be also recorded at 1, 3, 5 and 7 mm from the bone crest. If there is any discrepancy between buccal and lingual bone crest, the most apical one will be chosen as the reference.

In order to assess changes in bone crest height, the distance between the most coronal point of the bone crest (buccal and lingual) and the reference line tangent to a fixed reference point was calculated in mm.

BPT and RW at 1, 3, 5 and 7 mm will be also assessed when the implant has been already explanted, recording the months that have passed from the explantation.

For the characterization of the peri-implantitis defects, the defect morphology and severity classification by Monje and coworkers will be followed (Monje et al. 2019):

* Morphology:

  * Class I: Infraosseous defect. Class Ia: Buccal dehiscence. Class Ib: 2-3 walls defect. Class Ic: Circumferential defect.
  * Class II: Supracrestal/horizontal defect.
  * Class III: Combined defect. Class IIIa: Buccal dehiscence + horizontal bone loss. Class IIIb: 2-3 walls defect + horizontal bone loss. Class IIIc: Circumferential defect + horizontal bone loss.
* Severity: based upon the defect depth from the implant neck and ratio of bone loss/total implant length

  * Grade S: Slight: 3-4 mm/<25% of the implant length
  * Grade M: Moderate 4-5 mm/ ≥25%-50% of the implant length
  * Grade A: Advanced: >6 mm/>50% of the implant length

Regarding the statistical analysis, the statistical package (SPSS 15.0, SPSS Inc., Chicago, IL, USA, STATISTICS, version 7.1StatSoft, Inc. will be used for this purpose. The Pearson correlation test will be applied for the assessment of confounding factors and Linear regression models based on generalized estimating equations (GEEs) will be used to analyze the differences in the mean values of the post-extraction bone changes during the 2 time phases. This model will consider the correlations of within-subject repeated measures.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18-80 years
* patients with partial or complete edentulism with ≥1 missing teeth restored with implant-supported restorations
* patients with implants which had been in function for a minimum of 36 months after final prosthesis delivery
* patients presenting implant explantation due to peri-implantitis

Exclusion Criteria:

* pregnancy or lactation patients
* patients treated by zygomatic or pterygoid implants
* patients under intake of medications known to modify bone metabolism
* patients with uncontrolled systemic diseases (ie: diabetes mellitus)
* patients with active periodontal disease that required treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient recruitment will be obtained from a private practice exclusively dedicated to periodontics and implantology (Clinica CICOM, Badajoz, Spain). Edentulous patients, either total or partial, who previously underwent implant placement procedure and which suffer severe peri-implantitis will be consecutively included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2020-08-15 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
bone level changes | 4-6 months after implant explantation
  bone level changes (mm) and peri-implant defect morphology alterations after implant explantation

CONTACTS AND LOCATIONS:
Overall Officials: Jose Nart, Study Chair — Universitat Internacional de Catalunya
Locations (1):
- Universitat Internacional de Catalunya, Sant Cugat del Vallès, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pons R, Carreno M, Amerio E, Gargallo-Albiol J, Nart J, Monje A. Hard tissue dimensional changes following implant removal due to peri-implantitis: A retrospective study. Clin Implant Dent Relat Res. 2021 Jun;23(3):432-443. doi: 10.1111/cid.13004. Epub 2021 May 4. PMID 33949080